CLINICAL TRIAL: NCT04908644
Title: Study to Evaluate Efficacy and Safety of MS 20 on Patients With Ulcerative Colitis
Brief Title: MS-20 on Patients With Ulcerative Colitis(UC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202006118MIPB; MB103CLAS07 (Other: protocol No.)
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; MS-20; Postbiotics; Gut microbiota
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS-20 oral solution (Experimental): Oral Solution 8 c.c per day divided twice daily (BID) for 12 weeks.
  Interventions: Drug: MS-20 oral solution
- Placebo (Placebo Comparator): Oral Solution 8 c.c per day divided twice daily (BID) for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MS-20 oral solution — Fermented soybean extract MicrSoy-20(MS-20), which uses a variety of lactic acid bacteria and yeasts to metabolize organic soybeans
  Other Names: Chemo young
  Arms: MS-20 oral solution
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a small pilot study of the fermented soybean extract MicrSoy-20(MS-20) to confirm its ability to improve UC severity with the treatment of standard therapies.

The primary endpoint, structural alteration of gut microbiota during the trial will be analyzed. Secondary endpoints aim to observe the changes of partial Mayo score, patient response of medication of UC treatments, biomarker changes in blood, and safety after taking MS-20.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged between 20 and 65 years old who has confirmed diagnosis of moderate to severe Ulcerative Colitis (UC): partial Mayo score≧3.
2. Subject has established diagnosis of ulcerative colitis for≧3 months prior to screening.
3. Females with childbearing potential must agree to completely abstain from sexual intercourse or use adequate contraceptive methods such as IUD or birth control pills during the trial period. [Definition of infertility: (1) Menopause for at least 1 year; (2) Has undergone surgical ligation, such as hysterectomy, bilateral oophorectomy, or fallopian tube ligation; (3) Congenital structural abnormalities.
4. As judged by the investigators, subject who is proactive, have the ability to communicate with study staff, and capable and willing to cooperate two points below,

   1. be willing and able to comply with the subject visit arrangements and procedures defined in the protocol.
   2. to collect, store with adequate refrigerating facilities and delivery of stool samples from home.

Exclusion Criteria:

1. Subject who is allergic to soybean and its products.
2. Subject who has a history of human immunodeficiency virus (HIV) infection. (Through oral disclosure and medical records by the doctor, subject who decline to disclose will be excluded)
3. Subject cannot take drugs orally or have any gastrointestinal history or surgery which investigator believes may affect the absorption of the oral investigational product.
4. Subject who has known history of Crohn's disease
5. Subject who has used antibiotics, antifungal or antiviral drugs (not including skin topical medication) within 30 days before the screening visit.
6. Subject who has used probiotics and prebiotics-related products within 14 days before the screening visit (e.g., yogurt drink, yogurt, Yakult, Wakamoto tablets, Shin Biofermin S tablets, probiotic powder, fermented beverages, tablets, capsules, inulin, oligosaccharide products, etc.).
7. Subject who has used Chinese medicine or products containing such ingredients within 14 days before the screening visit.
8. Subject who had diarrhea caused by gastrointestinal infections within14 days before the screening visit (more than three soft or watery stools within 24 hours). Ulcerative colitis-induced diarrhea is unrestricted.
9. Woman who is pregnant, breastfeeding, or expect to breastfeed during the study period.
10. Subject who has any of the following abnormalities of biochemical lab results: AST or ALT (> 3 × upper limit of normal [ULN]) or higher; Total bilirubin ≥ 3 x ULN; Serum creatinine> 2 × ULN.
11. Subject who has a history of malignant tumors within five years before the screening visit, except for locally curable cancers that have been clearly cured, such as basal or squamous-cell carcinoma, superficial bladder cancer, or prostate, cervix, or breast carcinoma in situ.
12. The subject has a medical history of drug or alcohol addiction that may result in the inability to complete the trial at the investigator's discretion.
13. Subject who has participated in a clinical trial of other investigational drug treatments or medical devices within 30 days before the screening visit.
14. Subject who had Clostridium difficile infection.
15. Subject who has been abroad for more than 10 days in the 30 days before the screening visit or expected to go abroad for more than 10 days during the trial period.
16. The investigator judges that the subject is not suitable for participating in the trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline structural of gut microbiota at 16 weeks | Baseline, week 16
Change from baseline in the abundance and variability of gut microbiota at 16 weeks | Baseline, week 16

SECONDARY OUTCOMES:
Change from baseline of Partial Mayo Score at 12 weeks | Baseline, week 12
  Partial Mayo score consisted of 3 sub-scores: stool frequency, most severe rectal bleeding of the day, endoscopic findings and global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher scores indicated more severe disease.
Change from baseline of IL-6 level in blood at 12 weeks | Baseline, week 12
Change from baseline of TNF-α level in blood at 12 weeks | Baseline, week 12
Change from baseline of IL-1β level in blood at 12 weeks | Baseline, week 12
Change from baseline of IL-23 level in blood at 12 weeks | Baseline, week 12
Change from baseline of IL-33 level in blood at 12 weeks | Baseline, week 12
Change from baseline of C-reactive protein(CRP) level in blood at 12 weeks | Baseline, week 12
Change from baseline of erythrocyte sedimentation rate(ESR) at 12 weeks | Baseline, week 12
Change from baseline of fecal calprotectin result at 12 weeks | Baseline, week 12
Change from baseline of fecal occult blood result at 12 weeks | Baseline, week 12
Adverse events | up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan